CLINICAL TRIAL: NCT00005414
Title: Validation of a Historical Physical Activity Survey
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4332; R03HL047478 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To compare long-term recall of physical activity up to 15 years in the past with physical activity reports and physical fitness levels assessed at the baseline examination.

DETAILED DESCRIPTION:
BACKGROUND:

Sedentary habits in middle-aged individuals are associated with increased risk for cardiovascular disease. Studies examining this association typically have assessed physical activity participation in a narrow window, (for example, 1 week or 1 month) relative to probable disease etiology and progression. When the study was initiated, the possible relation of long-term physical activity patterns over decades or a lifetime to disease risk was not known because there existed no validated method of determining such exposure, but such studies were needed. It was hypothesized that validation of long-term recall of activity could lead to the application of lifetime physical activity patterns questionnaires. Data on lifetime activity patterns might be useful in case-comparison and prospective studies of cardiovascular disease.

DESIGN NARRATIVE:

Data analyzed for this project were from a cohort that had been under observation in the Aerobics Center Longitudinal Study. Baseline preventive medical examinations were given to 6,902 men and women during the interval from 1971-1982. Current physical activity and physical fitness levels (maximal exercise treadmill test) were assessed at baseline. Participants also completed a lifetime physical activity pattern questionnaire as part of a mail survey done in 1986. Self-reported physical activity from the 1986 questionnaire was used to categorize participants' physical activity levels for the years 1971-1985. These recalled levels of activity were compared to physical activity and physical fitness levels assessed during those same years at the baseline examinations (measure of truth). For example, participants who reported in the 1986 survey that they engaged in relatively high levels of physical activity in 1976 were expected to have recorded higher levels of physical fitness at the 1976 examination than participants who reported in 1986 that they were relatively sedentary in 1976. The study design permitted evaluation of how accurately participants recalled their physical activity up to 15 years in the past and allowed quantification of the errors investigators might expect from such assessments.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Study Completion 1993-09 (Actual)